CLINICAL TRIAL: NCT07339735
Title: A Phase 1, Open-Label Study to Assess the Relative Bioavailability of Two LY4064809 Formulations in Healthy Adult Participants
Brief Title: A Study of LY4064809 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 27796; J6M-MC-JSGG (Other: Eli Lilly and Company)
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — STX-478

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY4064809 Test (Experimental): LY4064809 test (Phase 3 formulation) formulation administered orally in one of two periods.
  Interventions: Drug: LY4064809 Test Formulation; Drug: LY4064809 Reference Formulation
- LY4064809 Reference (Experimental): LY4064809 reference (Phase 1 formulation) formulation administered orally in one of two periods.
  Interventions: Drug: LY4064809 Test Formulation; Drug: LY4064809 Reference Formulation

INTERVENTIONS:
Drug: LY4064809 Test Formulation — Administered orally
  Other Names: STX-478
Drug: LY4064809 Reference Formulation — Administered orally
  Other Names: STX-478

SUMMARY:
The purpose of this study is to find out how much LY4064809 gets into the blood stream and how long it takes the body to get rid of it when it is given as two formulations. For each participant, the study will last about nine weeks. Participants will remain in the clinical research center for about one month.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy as determined by medical evaluation, including medical history, physical examination, vital signs, and electrocardiogram (ECG) at screening and admission.
* Have clinical laboratory test results within the normal range
* Have normal blood pressure and pulse rate or not clinically significant
* Have a BMI within the range 18 to 32 kg/m2
* Participants assigned male at birth or assigned female at birth who are not of childbearing potential

Exclusion Criteria:

* History or presence of any of the following conditions, deemed clinically significant by the investigator (or designee):

  * metabolic disease, including congenital non-hemolytic hyperbilirubinemia, for example, Gilbert syndrome
  * bile duct disease, including removal of the gall bladder
  * digestive system disease
  * blood disease
  * disease of the nervous system
  * significant history of, or presence of, liver disease, including any abnormal liver function tests
  * heart disease
* Have an abnormal electrocardiogram (ECG) at screening or admission
* History of a major surgical procedure within 30 days prior to screening
* Diagnosed or treated cancer within 5 years prior to screening, with the exception of the following cancers cured through treatment: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and in situ carcinoma of the cervix cured through surgery

  * Clinically significant history of multiple or severe drug hypersensitivity reactions or drug allergies, as determined by the investigator
* Have used or plan to use medication within 14 days prior to admission, or plan to use during the study with the exception of acetaminophen
* Have creatinine lab clearance less than 90mL/min calculated using the Cockroft-Gault equation at screening
* Have a positive Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody or human immunodeficiency virus 1 and 2 antibody results at the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY4064809 | Predose on Day 1 Through Day 28
  PK: Cmax of LY4064809
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4064809 | Predose on Day 1 Through Day 28
  PK: AUC of LY4064809

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Fortrea Clinical Research Unit Inc. - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No